CLINICAL TRIAL: NCT06258746
Title: A Clinical Study on Absorption, Metabolism, and Excretion of [14C]HSK31679 in Healthy Adult Male Chinese Subjects - Mass Balance and Biotransformation of [14C]HSK31679 in Human
Brief Title: Pharmacokinetics, Mass Balance, and Metabolism of [14C]HSK31679 in Healthy Adult Male Volunteers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xizang Haisco Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK31679-102
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 160 mg/100 μCi [14C]HSK31679 (Experimental): [14C]HSK31679
  Interventions: Drug: [14C]HSK31679

INTERVENTIONS:
Drug: [14C]HSK31679 — A single oral dose of 160 mg/100 μCi [14C]HSK31679 after fasting for at least 10 hours.

SUMMARY:
This is a single-center, nonrandomized, and open design study to investigate the pharmacokinetics, mass balance, metabolism and excretion of HSK31679 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, Age: 18~45 years old (inclusive);
2. A total body weight ≥50 kg and BMI of 19 to 26 kg/m^2(inclusive);
3. Subjects who are willing to sign an informed consent form, able to communicate with the investigator and to complete all trial procedures as per the protocol.

Exclusion Criteria:

1. Clinically significant abnormal results for comprehensive physical examination, vital signs, routine laboratory tests [blood routine, blood biochemistry, coagulation routine, urine routine, Fecal analysis, thyroid function and antibodies, visual acuity and ophthalmic examination (slit lamp, introcular pressure, and fundoscopy), 12-lead electrocardiogram (ECG), chest X-ray (anteriorposterior), and abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, and kidney);
2. Positive for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, or Treponema pallidum antibodies;
3. Use of any Western medicine or Chinese patent medicine (including prescription drug, over-the-counter drug, health care product, or live attenuated influenza vaccine) within 14 days prior to screening;
4. Participation in any clinical trial and interference with other investigational drug or medical device within 3 month prior to screening;
5. Any clinical serious illness that has previously or currently affected the cardiovascular system, digestive system, respiratory system, endocrine system, nervous system, hematology, immunology, skin, tumors, psychiatry, and metabolic abnormalities, or any other disease or physiological condition that can interfere with trial results;
6. Have undergone major surgery within 6 months prior to screening or with incomplete healing of the surgical incision; major surgery includes, but is not limited to, any surgery with significant risk of bleeding, prolonged general anesthesia, or incisional biopsy or obvious traumatic injury (excluding cured appendicitis surgery or rectal prolapse surgery);
7. Severe allergic constitution, including known allergy to THR- β receptor agonists or any excipient of this investigational product, two or more drugs and food components, or with special dietary requirements and thus unable to follow a standardized diet;
8. Concomitant hemorrhoids or perianal diseases with regular/ongoing rectal bleeding;
9. Subjects who had Irregular bowel movements or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
10. Excessive drinking or frequent drinking within the first 6 months of the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine); Positive alcohol breath test during the screening period;
11. Subjects who smoked more than 5 cigarettes a day or habitually used nicotine-containing products in the 3 months before the screening period and could not quit during the test period;
12. Drug abuse or dependence, urine screening positive for drug abuse;
13. Habitually drinking grapefruit juice or excessive (more than 8 cups a day, 1 cup =250mL) tea, grapefruit, coffee, drinks containing caffeine or grapefruit, and could not quit during the test period;
14. Subjects who need to work in a condition with long-term radioactive exposure; or who have experienced significant radioactive exposure (≥2 chest/abdominal CT scans, or ≥3 other types of X-rays) within 1 year or participated in the radiopharma labeling test prior to the test;
15. Subjects who have a birth plan during the study period and within 1 year after completion of the study, or who don't agree that the subject and his or her spouse should take strict contraceptive measures (condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.) during the study period and within 1 year after completion of the study;
16. Subjects who have experienced blood loss or donated 400 mL of blood within the first 3 months of the screening period, or have received blood transfusions within 1 month;
17. Volunteers judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 6 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mass balance | From the start of administration to 240 hours after administration
  Percentage of cumulative drug excretion of [14C]HSK31679 on biological pecimens(urine and faeces) accounting for total radiation drug dose

SECONDARY OUTCOMES:
AUC(0-t) | From the start of administration to 240 hours after administration
  The pharmacokinetic parameters of HSK31679 and major metabolites (if applicable) in plasma
AUC(0-∞) | From the start of administration to 240 hours after administration
  The pharmacokinetic parameters of HSK31679 and major metabolites (if applicable) in plasma
Cmax | From the start of administration to 240 hours after administration
  The pharmacokinetic parameters of HSK31679 and major metabolites (if applicable) in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China